CLINICAL TRIAL: NCT03433157
Title: Clinical and Radiological Evaluation of Stainless Stain Crowns (SSCs) Placed Using the Hall Technique and Traditional Technique
Brief Title: Assessment of Stainless Stain Crowns Placed Using the Hall Technique and Traditional Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zafer Cavit Cehreli, DDS, PhD, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hall vs SSC
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Primary Teeth; Dental Caries; Dentin, Carious
Keywords: stainless stain crowns; Hall technique; children
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hall technique (Experimental): SSCs placed on primary teeth using Hall technique
  Interventions: Device: Hall technique
- Traditional technique (Active Comparator): SSCs placed on primary teeth using Traditional technique
  Interventions: Device: Traditional technique

INTERVENTIONS:
Device: Hall technique — Metal Stainless stain crown placed with Hall technique
  Arms: Hall technique
Device: Traditional technique — Metal Stainless stain crown placed with Traditional technique
  Arms: Traditional technique

SUMMARY:
The purpose of this study is to evaluate and compare the clinical performance of Stainless Stain Crowns Placed Using the Hall Technique and Traditional Technique

DETAILED DESCRIPTION:
Stainless Stain Crowns (SSCs) will be placed on two primary molar teeth with proximal caries, in a split mouth design. 200 patients will be included in the study. The teeth will be randomized into two groups according to the technique.

Group 1: SSCs that will be placed using Traditional Technique Group 2: SSCs that will be placed using Hall Technique The cooperation of the child during the procedure will be assessed with Frankl scale. The crowns will be evaluated at baseline and 1., 6., 12., 18., 24. months. Radiographical evaluations will be at 6.,12. and 24. months. The data will be analysed statistically using chi square test and Log-Rank test and the Kaplan-Meier survival method will be used to estimate survival percentages.

ELIGIBILITY:
Inclusion Criteria:

* Patients and parents of the patients who accept to participate and sign the informed consent
* Patients who have two first and/or second primary molars with caries affecting at least two surfaces
* Patients who are cooperative for the dental procedure

Exclusion Criteria:

* Patients and parents of the patients who does not accept to participate and sign the informed consent
* Teeth that are previously restored
* Patients with a systemic disease,
* Patients who have orthodontic treatment
* Teeth which have a short period of time for succedaneous teeth to erupt
* Teeth which need vital or non-vital endodontic treatment
* Patients and/or parents who does not accept the esthetic appearance of SSC

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Clinical performance of Stainless Stain Crowns (SSCs) Placed Using the Hall Technique and Traditional Technique | 2 years
  Assessment of SSCs placed with two different techniques on primary molar teeth. The cooperation of children will be assessed with Frankl Scale (1:definitely negative, 2:negative, 3:positive, 4:definitely positive).
  Evaluation criteria will be;
  * spontaneous pain (absent/present);
  * tenderness to percussion/palpation (absent/present);
  * mobility (no mobility/ 1mm/ 2mm/ 3mm mobility)
  * swelling (absent/present);
  * fistula (absent/present)
  * periapical/interradicular radiolucency (absent/present);
  * widened periodontal ligament (absent/present);
  * loss of lamina dura (absent/present);
  * internal/external root resorption (absent/present)
  * the marginal adaptation of each crown: good when the margins were sealed / poor when the margins were open
  * retention of the crown (absent/ present)
  * fracture of the crown (absent/ present)
  * gingival health/gingivitis (absent/ present)
  * plaque around the crown (absent/ present)

CONTACTS AND LOCATIONS:
Overall Officials: Zafer C Cehreli, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Innes NP, Stewart M. The Hall Technique, a Simplified Method for Placing Stainless Steel Crowns on Primary Molars, may be as Successful as Traditionally Placed Crowns. J Evid Based Dent Pract. 2015 Jun;15(2):70-2. doi: 10.1016/j.jebdp.2015.03.008. Epub 2015 Mar 28. No abstract available. PMID 25987388